CLINICAL TRIAL: NCT05262920
Title: Promoting Self-Management of Breast and Nipple Pain With Technology (PROMPT) for Breastfeeding Women Study
Acronym: PROMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Hartford HealthCare (Other); UConn Health (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ruth Lucas, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E21-0205; R56NR020041 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-03-02 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding, Exclusive; Pain, Acute; Maternal Distress; Parent-Child Relations; Self Efficacy
Keywords: Breastfeeding, Pain, Self-efficacy
MeSH Terms: conditions — Breast Feeding; Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: The proposed Randomized Control Trial (RCT),will be conducted to test the effect of the BSM intervention vs. an attention control group on BNP, BF exclusivity and duration, BF self-efficacy, and maternal well-being to 24 weeks
Who Masked: Participant, Investigator
Masking Description: The investigators will employ blinding whenever possible. The investigators team members involved in data collection or analysis will be blinded to the group assignment of participants. Research team personnel will follow a strict script to refrain from discussing participant activities, and by using the data management graduate assistant (unblinded) to coordinate assigned condition activities and data collection and analysis. All participants will be assigned a study number, which will be used to track the study measures. De-identified data with dummy codes for assigned condition will be entered into the study database to allow blinded data analysis. Blinding was successfully employed during the BSM pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The BSM Intervention (Experimental): Guided by the Individual and Family Self-Management Theory, the Lucas team developed the Breastfeeding and BNP Self-Management (BSM) intervention. The BSM intervention uses a cloud-based platform, links to educational modules, and daily journaling, to provide women uniform best practice knowledge and skills for BF and BNP self-management.
  Strategies include guided imagery, therapeutic breathing, mindfulness, relaxation, non-pharmacological interventions that are integrated within the self-management process such as goal-setting, self-monitoring, problem-solving, and social support through texting.
  Interventions: Behavioral: The BSM Intervention
- Attention Control (Active Comparator): Attention control participants will receive equivalent attention as the BSM group. The fourth-trimester care based on the Centers for Disease Control (CDC) HEAR HER campaign and infant health information modules will be provided through the REDCap link.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: The BSM Intervention — The BSM intervention entailed a daily electronic journal for monitoring BF and BNP with feedings, bi-weekly texting for 6 weeks from a research nurse for informational support and to promote personalized goal-setting and problem-solving, and hyperlinks to eight uniform BNP educational modules (knowledge and skills) and online resources. 1. Fundamentals of BF (FBF), 2. Deep breathing (DB), 3. BNP non-pharmacological strategies (BNPS), 4. Guided imagery (GI), 5. Pain neurophysiology specifically related to BF (PN-BF), 6. Catastrophizing, 7. Stress reactivity, and 8. Common pumping issues and interventions (CPI).
  Arms: The BSM Intervention
Behavioral: Attention Control — The Attention Control and Intervention groups both receive fourth-trimester care videos. The educational modules are the following: Urgent maternal warning signs, caring for the maternal body after birth; infant care; Coronavirus disease 2019 (COVID-19) and infant health prevention; maternal and infant immunization; infant safety in the home; maternal and infant dietary recommendations; and national and health resources to support BF in the workplace
  Arms: Attention Control

SUMMARY:
Every year, 1 million women cease breastfeeding (BF) before 6 months, the minimum time required for optimal maternal and infant health, development, and well-being. The highest rate of BF cessation occurs within 3 weeks after birth, with 30% of women ceasing BF due to acute breast and nipple pain (BNP). BNP is a complex and understudied biobehavioral phenomenon involving nociceptive signaling that stimulates multiple pain pathways. Women who experience BNP beyond BF initiation report lower BF self-efficacy, a key predictor of BF at 6 months and increased maternal distress symptoms contributing to differences in early BF cessation rates. The investigators developed and tested their 6-week nurse-led and participant-informed, Breastfeeding and Breast and Nipple Pain Self-Management (BSM) intervention guided by the Individual and Family Self-Management Theory. Aligned with the needs and preferences elicited from BF participants, the investigators used a cloud-based platform to deliver BF knowledge and skills and provided support through nurse-led text-based communication to decrease BNP, increase BF self-efficacy, decrease burdensome face-to-face visits, and increase adaptive coping behaviors. Participants in the BSM intervention group reported significantly reduced BNP intensity at 1 and 2 weeks which predicted increased BF self-efficacy and decreased anxiety at 6 weeks. Based on these promising results, the investigators propose to examine the efficacy of the BSM intervention in an R56NR020041 Randomized Control Trial (RCT), Promoting Self-Management of Breast and Nipple Pain Using Technology (PROMPT) for Breastfeeding Women to decrease BNP intensity and interference and increase BF exclusivity. The study will reproduce and extend the pilot findings by exploring in a diverse population of BF participants how participants' pain sensitivity affects BNP. The study will explore the moderating role of BNP, and maternal well-being symptoms of fatigue, depressive symptoms, anxiety, and sleep, pain, pain coping, and maternal self-efficacy, on BF exclusivity. Participants (N = 222) intending to breastfeed will be randomized to the BSM intervention or the attention control group with assessments performed at baseline, 1, 2, 3, 6, 9, 12, 18, and 24 weeks. Study results will advance knowledge on the BSM intervention, with direct implications for nurse-designed and lead self-management interventions in clinical settings or health care systems.

DETAILED DESCRIPTION:
In response to the critical gap that exists in identifying effective biobehavioral self-management interventions for participants during BF initiation who experience breast and nipple pain (BNP), the investigators developed a patient-informed Breastfeeding and BNP Self-Management (BSM) intervention based on the Individual and Family Self-Management Theory. The investigators propose to test the effectiveness of the BSM intervention on BNP severity, pain interference with daily life, and BF outcomes over time in this R56NR020041 Randomized Control Trial, Promoting Self-Management of Breast and Nipple Pain with Technology (PROMPT) for Breastfeeding Women. Participants (N=222) intending to BF will be randomized either to receive the BSM intervention or be in the attention control group, with assessments performed after birth at the hospital (baseline). After screening and informed consent, participants will be asked to complete study measures, undergo quantitative sensory testing using a standardized protocol, and access a secure electronic survey site via participants' smartphone or study-provided smartphone text links or email before discharge home. During the first week home, all participants will receive bi-weekly texts with links to BSM intervention BF modules or for the attention control group, educational modules on postpartum recovery and infant care. All participants at 1, 2, 3, 9, 12, and 18 weeks will receive a text or email for ongoing assessments of BNP and BF measures of the exclusivity (breast, breast milk, or formula), the number of feedings each day, and how long (days/weeks/months) infants were breastfed (duration). In addition, the study occurs via mobile technology during an acute period of pain when the rate of BF cessation is the highest. At 6- and 24-weeks participants will repeat the study measures and quantitative sensory testing.

The PROMPT study is the first to target self-management for BNP using cloud-based educational modules and user-preferred text-based smartphone intervention during the critical weeks of BF initiation, when support for BF is most desired, face-to-face visits are most burdensome, and places the mother-infant dyads at risk for illness, such as COVID-19. The study will describe how many participants experience BNP from BF initiation to 24 weeks as participants return to work and who may be at risk for chronic pain, which has not been examined. The study also replicates and expands on how the presence of pain sensitivity affects BNP and BF outcomes. The results from this study hold great promise to 1) support a diverse population of BF participants by identifying the risk factors of BNP; 2) target personal interventions for participants experiencing BNP based on unique moderating factors of pain sensitivity, nonpharmacological interventions, BF self-efficacy, pain coping, maternal self-efficacy and maternal well-being (anxiety, depression, stress, and fatigue); and 3) to develop easily accessible strategies for participants BF within clinical settings that allow for large-scale translation in health care systems or public health settings.

Participant Recruitment will begin by active and passive methods successfully used in the pilot study with the addition of prenatal recruitment in the clinical site. Passive methods include (1) advertisements via Facebook pages (Connecticut Breastfeeding Coalition and the School of Nursing Center for the Advancement of Management of Pain (CAMP)) and Instagram ads, targeting participants in Connecticut who intend to BF, (2) flyers posted at clinical partners offices, (3) flyers given by the clinical partners to participants expressing interest in BF during routine prenatal care and referring participants to the peer counselors, research assistants, or lactation consultants team members on the inpatient hospital units, (4) flyers included in discharge educational packets at both recruitment sites, (5) flyers posted in hospital (HH, University of Connecticut Medical Center (UConn Health) common areas.

Active methods include screening the inpatient unit census two to three times per week by the clinical partners for participants who meet inclusion or exclusion criteria. Participants who agree to speak with a member of the research team about the study will be approached. A HIPAA consent will be obtained for the research team to ask initial screening questions via REDCap (Research Electronic Data Capture). REDCap is a secure web application and database storage for creating and managing online data collection with highly customizable data types (including 21 Code of Federal Regulations (CFR) Title 21 Part 11, Federal Information Security Modernization Act (FISMA), and Health Insurance Portability and Accountability Act (HIPAA) compliant environments). If eligible, informed consent will be obtained by a member of the research team trained in obtaining informed consent and approved by the Institutional Review Board (IRB).

The investigators will recruit participants after birth, with data collection to occur before discharge from the hospital and take approximately 60 minutes. To decrease participant burden, recruitment will begin during the antenatal care so participants may anticipate participating in data collection after delivery. In BSM pilot study, the retention rate was 94% of participants at 6 weeks, and as the primary aim is the effectiveness of the intervention during the first 3 weeks, the sample size calculations account for the possibility of loss-to-follow-up as high as 5% at 3 weeks. Additionally, the investigators anticipate the possibility of a 25% attrition rate at 24 weeks, a level somewhat larger than the 15-20% rate observed in many longitudinal intervention trials.

After informed consent and prior to the start of data collection, participants will be randomized to the BSM intervention or the attention control group and be assigned a unique participant identification number. Participants will be shown how to access the REDCap modules on participants' or a study-provided smartphone. An alternative contact person's information will be requested to reduce the likelihood of attrition. A randomization schedule created in REDCap will ensure that the two groups remain balanced with respect to age, race, BF experience, antenatal plan for BF duration, route of delivery, and intent to return to work. The randomization assignment will be known to data management graduate assistant with experience in clinical trials, intervention monitoring, IRB compliance. The PI will be blinded to the randomization assignment of participants. The graduate assistant will not be involved in data collection but will administer and monitor the interventions and missing data.

After discharge, both groups will receive an encrypted text via REDCap with embedded links from Twilio, a cloud communications platform, and a backup archive feature to secure participant's privacy and confidentiality, from the nurse on the research team. The follow-up measures at 1, 2, 3, 9, 12, and 18 weeks (Figure 4, see research plan) include the participants weekly BNP, pain coping, BF exclusivity, ongoing BF assessment, BF algorithm, and maternal assessment of infant BF behaviors, self-efficacy scales (pain, BF, and maternal), maternal well-being assessments, and perceived well-being scales. The completion of the measures will take about 30 minutes. Weekly meetings will identify any missing data and contact participants to complete the surveys. At 6 and 24 weeks, participants will complete the above measures and quantitative sensory testing at the clinical locations. The completion of the measures will take about 60 minutes.

Intervention Administration. Each group will receive a link to the eight video modules that address a different topic within a 15-minute interval. During the first week, the appropriate link to the first video to the BSM intervention and attention control group will be sent. Intervention fidelity will be addressed using continual assessment of design, training, delivery, receipt, enactment throughout the study duration. Design fidelity is applied through a standardized intervention with scheduled interactive texts, text-based daily BF journals and links to modules. Dr. Lucas will routinely assess the training of the interventionist(s) through simulated scenarios and practice sessions using texting and phone scripts. Evidence of treatment will include participant's response to bi-weekly texts and targeted lactation support based on galactogenesis and lactation milestones. The investigation team will monitor intervention fidelity by using the REDCap feature that allows the study team to view the date, time, length, and the number of times the participant accesses each module and completes the daily BF journal. The Project Manager will coordinate the study team to send participants text and follow-up phone calls at 1, 2, 3, 9, 12, and 18 weeks at a prescheduled time to encourage completion of the modules and for BSM intervention, address any BF concerns. After the first week, phone calls and encrypted text messages, depending on the participant preference, will be made by the research team to encourage BF data completion.

Participant Retention At enrollment, participants will be informed that payment will occur after each data collection point completion and if all data points are completed will receive a study completion bonus. To maintain contact and trust, the participants in both groups will receive monthly text links at 4, 8, 12, 16, 20, and 24 weeks, to modules highlighting normal infant development and age-appropriate play.

The sample size objective for the study is to recruit N = 222 participants who will be randomly assigned to the BSM or attention control study groups at a 1:1 ratio (111 per group). This objective provides 80 percent power (α =0.05, two-sided) to detect a standardized mean difference (Cohens d) of 0.39 or more between the BSM and attention control groups. It also provides 80 percent power to detect an odds ratio of 2.5 or more in exclusive BF between the two groups, assuming that the exclusive BF rate of the control group will be 10 percent higher than the national population rate in 2017 at 6, 9, 12, 18, and 24 weeks. These calculations account for "loss to follow-up" as high as 5% at 3 weeks and 25% at 24 weeks. The calculations reflect a conservative approach relative to the attrition rate of 6% that occurred at the 6-week time point in the pilot study and the 15-20% rate observed in many longitudinal intervention trials. In the pilot study, repeated measures ANCOVAs (with the baseline value of a measure as the covariate) revealed standardized mean differences larger than d = 0.39 for the main effect of the intervention on BNP intensity (d = 0.45), pain severity (d = 0.60), cumulative pain (d = 0.64), and BF self-efficacy (d = 0.48) cross the 1, 2, and 6 week time points. For BNP interference, the value of d was 0.39 at week 1, but smaller at weeks 2 and 6. Furthermore, the odds of exclusive BF in the intervention group is 2.9 times higher than the control group at 6 weeks, which is also higher than the hypothesized OR = 2.5. Therefore, the investigators are confident that the sample size goal will be sufficiently powered to detect intervention effects on key variables for study aims 1 and 2.

Finally, the sample size estimate does not reflect the investigators' plans to conduct analyses based on repeated measurement of outcome variables at the 1, 2, 3, 6, 9, 12, 18, and 24 week time points (due to the dearth of information regarding 24-week outcomes). Generally, the inclusion of data for an outcome variable across additional time points marginally enhances statistical power, especially for testing main and interaction effects of intervention and time.

ELIGIBILITY:
Please reformat the Eligibility Criteria. The preferred format includes lists of inclusion and exclusion criteria as shown below.

Inclusion Criteria:

* women
* 18 - 45 years of age
* Gave birth < 48 hours to a singleton infant > 37 weeks gestational age
* Intend to BF
* Received standardized BF basics during their antenatal care
* Access to the internet via own smartphone or study provided smartphone
* Able to read and write English
* Assessed by lactation consultant during BF

Exclusion Criteria:

* < 18 or > 45 years of age
* History of significant mental health disorder (e.g., major depression, schizophrenia, or bipolar disorder) due to additional challenges in the capacity for self-management
* Skin conditions on nondominant forearm which could interfere with quantitative sensory testing
* Birth of an infant with medical complications or congenital anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female able to directly breastfeed. Males and transgender males at this time are unable to BF and not eligible for this study.
Enrollment: 250 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth F Lucas, PhD, Principal Investigator — University of Connecticut
Locations (2):
- United States (2):
  - UConn Health, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
The final research data will be a computerized dataset consisting of participant data, BF exclusivity, BNP, and pain sensitivity. All data will be shared and published in a de-identified manner and free of identifiers that would permit linkages or variables that may lead to deductive disclosure of the identity of the individual participants.
  Data generated from the proposed study will be shared with and available to the participating study investigators. We also intend to make results available upon request to the community of scientists interested in BF and BNP.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Datasets will also be shared with other qualified researchers after major publications have been accepted which will be 5 years after the study is completed.
Access Criteria: Datasets will be made readily available for sharing across the maternal child and BF research groups at the UConn. Furthermore, we will welcome collaboration with maternal child clinicians and others who may make use of the study protocols developed in the proposed study.

REFERENCES:
- [Background] Lucas RF, McGrath JM. Clinical assessment and management of breastfeeding pain. Top Pain Manag. 2016;32(3):1-12.
- [Background] Lucas R, Bernier K, Perry M, Evans H, Ramesh D, Young E, Walsh S, Starkweather A. Promoting self-management of breast and nipple pain in breastfeeding women: Protocol of a pilot randomized controlled trial. Res Nurs Health. 2019 Jun;42(3):176-188. doi: 10.1002/nur.21938. Epub 2019 Mar 5. PMID 30835887
- [Background] Lucas R, Zhang Y, Walsh SJ, Evans H, Young E, Starkweather A. Efficacy of a Breastfeeding Pain Self-Management Intervention: A Pilot Randomized Controlled Trial. Nurs Res. 2019 Mar/Apr;68(2):E1-E10. doi: 10.1097/NNR.0000000000000336. PMID 30829925
- [Background] Gallegos D, Russell-Bennett R, Previte J, Parkinson J. Can a text message a week improve breastfeeding? BMC Pregnancy Childbirth. 2014 Nov 6;14:374. doi: 10.1186/s12884-014-0374-2. PMID 25369808
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Subnis UB, Starkweather A, Menzies V. A current review of distraction-based interventions for chronic pain management. Eur J Integr Med. 2016;8(5):715-722. doi:10.1016/j.eujim.2016.08.162
- [Background] Litt MD, Tennen H. What are the most effective coping strategies for managing chronic pain? Pain Manag. 2015;5(6):403-6. doi: 10.2217/pmt.15.45. Epub 2015 Sep 24. No abstract available. PMID 26399377
- [Derived] Aderibigbe T, Kelleher SL, Henderson WA, Prescott S, Young EE, Lucas RF. COMT Variants are Associated With Breast and Nipple Pain. J Pain. 2024 Sep;25(9):104568. doi: 10.1016/j.jpain.2024.104568. Epub 2024 May 18. PMID 38763257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began March 2022 and completed in June 2023. The recruitment sites were two academic medical centers maternity units.
Pre-assignment Details: Two participants were screened and were excluded from the study. All other participants were screened and enrolled in the study.
Groups:
- The BSM Intervention: Guided by the Individual and Family Self-Management Theory, the Lucas team developed the Breastfeeding and BNP Self-Management (BSM) intervention. The BSM intervention uses a cloud-based platform, links to educational modules, and daily journaling, to provide women uniform best practice knowledge and skills for BF and BNP self-management.
  Strategies include guided imagery, therapeutic breathing, mindfulness, relaxation, non-pharmacological interventions that are integrated within the self-management process such as goal-setting, self-monitoring, problem-solving, and social support through texting.
  The BSM Intervention: The BSM intervention entailed a daily electronic journal for monitoring BF and BNP with feedings, bi-weekly texting for 6 weeks from a research nurse for informational support and to promote personalized goal-setting and problem-solving, and hyperlinks to eight uniform BNP educational modules (knowledge and skills) and online resources. 1. Fundamentals of BF (FBF), 2. Deep breathing (DB), 3. BNP non-pharmacological strategies (BNPS), 4. Guided imagery (GI), 5. Pain neurophysiology specifically related to BF (PN-BF), 6. Catastrophizing, 7. Stress reactivity, and 8. Common pumping issues and interventions (CPI).
- Attention Control: Attention control (AC) participants will receive equivalent attention as the BSM group. The fourth-trimester care based on the Centers for Disease Control (CDC) HEAR HER campaign and infant health information modules will be provided through the REDCap link.
  Attention Control: The Attention Control and Intervention groups both receive fourth-trimester care videos. The educational modules are the following: Urgent maternal warning signs, caring for the maternal body after birth; infant care; COVID-19 and infant health prevention; maternal and infant immunization; infant safety in the home; maternal and infant dietary recommendations; and national and health resources to support BF in the workplace
Period: Overall Study
Arm/Group | The BSM Intervention | Attention Control
Started | 122 | 128
Completed | 77 | 97
Not Completed | 45 | 31

BASELINE CHARACTERISTICS:
Population: The study successfully recruited our target sample size of 222 in May 2023 and recruited an additional 28 women in June 2023, for a total of 250 participants (113%).
Groups:
- Attention Control: Attention control participants will receive equivalent attention as the BSM group. The fourth-trimester care based on the CDC HEAR HER campaign and infant health information modules will be provided through the REDCap link.
  Attention Control: The Attention Control and Intervention groups both receive fourth-trimester care videos. The educational modules are the following: Urgent maternal warning signs, caring for the maternal body after birth; infant care; COVID-19 and infant health prevention; maternal and infant immunization; infant safety in the home; maternal and infant dietary recommendations; and national and health resources to support BF in the workplace
- Total: Total of all reporting groups
Arm/Group | The BSM Intervention | Attention Control | Total
Number analyzed (Participants) | 122 | 128 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.16 (4.63) | 30.32 (5.19) | 30.24 (4.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 128 | 250
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 36 | 71
  Not Hispanic or Latino | 87 | 92 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 29 | 27 | 56
  White | 74 | 85 | 159
  More than one race | 11 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122 | 128 | 250
Visual Analogue Scale for Breast and Nipple Pain Severity [Mean (Standard Deviation); unit: units on a scale] — Visual analogue scale (0-100) uses an unlabeled line with scores further to the right indicating higher scores and increased pain The scale was collected via text-linked via REDCap
  units on a scale | 36.55 (25.05) | 39.43 (25.28) | 38.03 (25.16)
Brief Pain Inventory (BPI) Pain Intensity Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory (BPI) Pain Intensity sum score of 4 items (3, 4, 5, and 6). Each item is scored 0-10, the BPI pain intensity sum score ranges from 0-40. The higher the score the worse the pain. A composite score of the average is sometimes reported. Factor analysis verified the two separate factors, pain intensity and interference, found in the previous study. Internal stability (Cronbach alpha) was also examined in this study. Alphas showed good internal consistency, ranging from 0.80 to 0.87 for the four pain intensity items.
  units on a scale | 3.88 (1.96) | 3.79 (2.04) | 3.83 (2.00)
Brief Pain Inventory (BPI) Interference Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory pain interference is the average sum score of 7 items 9a - 9g. Each item is scored 0-5, with a total score of 0-35. Higher scores mean worse pain. A composite score of the average is sometimes reported. Factor analysis verified the two separate factors, pain severity and interference, found in the previous study. Internal stability (Cronbach alpha) was also examined in this study. Alphas showed good internal consistency, ranging from 0.89 to 0.92 for the seven interference item.
  units on a scale | 3.38 (2.4) | 3.55 (2.54) | 3.46 (2.47)
Breastfeeding Exclusivity Participation Rate [Count of Participants; unit: Participants] — The number of participants who self-reported breastfeeding exclusivity (providing only breast milk and no formula) their infant
  Participants | 119 | 118 | 237
Breastfeeding Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — Breastfeeding Self-Efficacy Scale is a 14 item scale with 5-point Likert scale (1-5). Score Range: 14-70, with higher scores (>50) indicate greater breastfeeding self-efficacy.
  units on a scale | 45.28 (13.71) | 45.49 (13.01) | 45.38 (13.36)
Anxiety Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form 6a [Mean (Standard Deviation); unit: t-score] — The PROMIS Short Form v1.0 - Anxiety 6a is a 6-item Likert Scale (1-5, never - always). Total raw score ranges from 6-30. Raw scores are converted to a T-score. The T-score of 50 is the population mean and the average for the US population with a standard deviation of 10. The T-score of 60 is indicative elevated levels of anxiety. PROMIS Anxiety shows moderate to strong correlations with Generalized Anxiety Disorder 7-item scale and Hospital Anxiety and Depression Scale-Anxiety.
  t-score | 51.56 (9.1) | 51.27 (8.37) | 51.41 (8.73)
Edinburgh Postnatal Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Edinburgh Postnatal Depression Scale is a 10-item questionnaire with a 0-3 Likert scale. The total score ranges from 0 to 30. A score of 10 or more may indicate possible depression and a score of 13 or higher may be used to identify women with higher risk for depression diagnosis.
  units on a scale | 5.56 (4.62) | 6.03 (4.92) | 5.79 (4.77)
Fatigue Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form 6a [Mean (Standard Deviation); unit: T-score] — The PROMIS Short Form v1.0 - Fatigue 6a is a 6-item Likert Scale (1-5, never - always). Total raw score ranges from 6-30. Raw scores are converted to a T-score. The T-score of 50 is the population mean and the average for the US population with a standard deviation of 10. The T-score of 60 is indicative of elevated levels of fatigue.
  T-score | 53.99 (9.63) | 54.95 (9.26) | 54.47 (9.44)
Perceived Stress Scale10 Form V.09/16/13 [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale (PSS-10) is a 10-item questionnaire is a 10-item Likert Scale from 0 ("Never") to 4 ("Very Often"). The total scores ranges from 0-40. To calculate a total PSS score, responses to the four positively stated items (items 4, 5, 7 and 8) first need to be reversed (i.e. 0 => 4; 1 => 3; 2 => 2; 3 => 1; 4 => 0). Higher scores indicate higher levels of perceived stress.
  units on a scale | 12.94 (6.66) | 12.93 (6.15) | 12.93 (6.40)
Sleep Disturbance Patient-Reported Outcomes Measurement Information (PROMIS) Short Form v1.0 - 6a [Mean (Standard Deviation); unit: T-score] — The PROMIS Short Form v1.0 - Sleep Disturbance 6a is a 6-item Likert Scale (1-5, never - always). Total raw score ranges from 6-30. Raw scores are converted to a T-score. The T-score of 50 is the population mean and the average for the US population with a standard deviation of 10. The T-score of 60 indicative of increased sleep disturbances.
  T-score | 52.35 (9.16) | 54.13 (9.09) | 53.22 (9.12)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale for Breast and Nipple Pain Severity
Description: Visual analogue scale (0-100) uses an unlabeled line with scores further to the right indicating higher scores and increased pain
Time Frame: Baseline to 24 weeks
Population: The visual analogue scale (0-100) will quantify breast and nipple pain severity during breastfeeding at all data points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control | The BSM Intervention
Number analyzed (Participants) | 128 | 122
units on a scale
  Baseline | 39.43 (25.28) | 36.55 (25.05)
  Week 1: number analyzed (Participants) | 116 | 108
  Week 1 | 44.31 (25.34) | 36.93 (27.61)
  Week 2: number analyzed (Participants) | 112 | 96
  Week 2 | 33.8 (26.26) | 25.68 (25.79)
  Week 3: number analyzed (Participants) | 107 | 94
  Week 3 | 31.42 (24.7) | 18.26 (21.19)
  Week 6: number analyzed (Participants) | 108 | 90
  Week 6 | 17.2 (22.1) | 8.86 (18.49)
  Week 9: number analyzed (Participants) | 99 | 81
  Week 9 | 12.21 (19.19) | 5.86 (14.86)
  Week 12: number analyzed (Participants) | 98 | 81
  Week 12 | 7.96 (14.53) | 6.22 (14.72)
  Week 18: number analyzed (Participants) | 93 | 73
  Week 18 | 4.33 (11.23) | 7.68 (17.52)
  Week 24: number analyzed (Participants) | 97 | 77
  Week 24 | 6.54 (13.75) | 5.75 (15.14)
Statistical Analysis 1: Comparison: Attention Control vs The BSM Intervention; Test type: Superiority; p < 0.0045, Genalized Linear Mixed Models
Statistical Analysis 2: Comparison: Attention Control vs The BSM Intervention; Test type: Superiority; p = 0.022, Generalized Linear Mixed Model

2. Primary Outcome: Brief Pain Inventory Pain Intensity Scale
Description: The Brief Pain Inventory pain intensity sum score of 4 items (3, 4, 5, and 6). Each item is scored 0-10, the pain intensity sum score ranges from 0-40. The higher the score the worse the pain. A composite score of the average is sometimes reported. Factor analysis verified the two separate factors, pain intensity and interference, found in the previous study. Internal stability (Cronbach alpha) was also examined in this study. Alphas showed good internal consistency, ranging from 0.80 to 0.87 for the four pain intensity items.
Time Frame: Baseline to 24 weeks
Population: The Brief Pain Inventory pain severity sum score (item 3, 4, 5, and 6) will quantify breast and nipple pain during breastfeeding at all data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
score on a scale
  Baseline | 3.88 (1.96) | 3.79 (2.04)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 3.56 (2.07) | 3.72 (1.81)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 2.89 (1.92) | 3.24 (1.92)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 2.52 (1.77) | 2.83 (1.89)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 2.38 (1.75) | 2.19 (1.56)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 2.00 (1.52) | 1.93 (1.46)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 1.64 (1.06) | 1.86 (1.44)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 1.89 (1.24) | 1.84 (1.42)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 1.81 (1.33) | 1.76 (1.19)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.65, Genalized Linear Mixed Models
Statistical Analysis 2: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.402, Generalized Linear Mixed Model

3. Primary Outcome: Brief Pain Inventory Interference Scale
Description: The Brief Pain Inventory Pain Interference score is the average sum score of 7 items 9a - 9g. Each item is scored 0-5, with a total score of 0-35. Higher scores mean worse pain. A composite score of the average is sometimes reported. Factor analysis verified the two separate factors, pain intensity and interference, found in the previous study. Internal stability (Cronbach alpha) was also examined in this study. Alphas showed good internal consistency, ranging from 0.89 to 0.92 for the seven interference item.
Time Frame: Baseline to 24 weeks.
Population: The Brief Pain Inventory pain interference sum score (items 9a - 9g) will quantify breast and nipple pain during breastfeeding effect on everyday life at all data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
score on a scale
  Baseline | 3.38 (2.40) | 3.55 (2.54)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 2.27 (2.34) | 2.46 (2.27)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 1.92 (2.47) | 2.00 (2.40)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 1.25 (2.06) | 1.36 (2.02)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 1.29 (2.42) | 1.11 (2.31)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 1.09 (2.42) | 0.95 (2.11)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 1.15 (2.7) | 0.89 (2.01)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 1.18 (2.60) | 0.63 (1.5)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 1.11 (2.47) | 0.92 (2.19)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.681, Generalized Linear Mixed Model
Statistical Analysis 2: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.529, Generalized Linear Mixed Model

4. Primary Outcome: Cumulative Breast and Nipple Pain Scores
Description: Each weekly score uses the visual analogue score of 0-100. Cumulative Breast and Nipple Pain (BNP) is calculated each week as a summed additive score. Participants' cumulative BNP (baseline +1 week, + 2 weeks, + 3 weeks, + 6 weeks, + 9 weeks, + 12 weeks, +18 weeks, 24 weeks, 0 - 900). Higher cumulative scores represent greater BNP severity.
  Only individuals who remain in the study scores are reported.
Time Frame: Baseline to 24 Weeks
Population: Participants reported BNP severity using a visual analogue scale (0 - 100) at baseline and across time. Participants' cumulative BNP (baseline, +1 week, + 2 weeks, +3 weeks, + 6 weeks, + 9 weeks, +12 weeks, +18 weeks, +24 weeks, 0 - 900)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
units on a scale
  Baseline | 36.55 (25.05) | 39.43 (25.28)
  1 Week: number analyzed (Participants) | 108 | 116
  1 Week | 72.47 (46.17) | 84.36 (45.1)
  2 Weeks: number analyzed (Participants) | 96 | 112
  2 Weeks | 98.57 (62.22) | 117.64 (63.76)
  3 Weeks: number analyzed (Participants) | 94 | 107
  3 Weeks | 115.63 (77.25) | 148.94 (80.14)
  6 Weeks: number analyzed (Participants) | 90 | 108
  6 Weeks | 126.59 (87.53) | 166.58 (92.43)
  9 Weeks: number analyzed (Participants) | 81 | 99
  9 Weeks | 132.32 (92.50) | 179.78 (104.46)
  12 Weeks: number analyzed (Participants) | 81 | 98
  12 Weeks | 141.54 (101.90) | 188.78 (111.35)
  18 Weeks: number analyzed (Participants) | 73 | 93
  18 Weeks | 150.85 (115.14) | 195.77 (114.62)
  24 Weeks: number analyzed (Participants) | 77 | 97
  24 Weeks | 160.37 (124.95) | 202.38 (122.25)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p < 0.011, MANOVA

5. Secondary Outcome: Breastfeeding Exclusivity Participation Rate
Description: The number of participants who self-reported breastfeeding exclusivity (providing only breast milk and no formula) their infant.
Time Frame: Baseline to 24 weeks
Population: Examine the effect of the BSM intervention on secondary outcomes of BF exclusivity. BF exclusivity is for the infant to receive only breast milk from the breast or bottle for al feeding.
Measure: Count of Participants; unit: Participants
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
Participants
  Baseline Exclusive Breastfeeding (EBF) | 119 | 118
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 67 | 74
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 56 | 70
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 50 | 57
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 48 | 61
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 43 | 61
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 43 | 58
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 37 | 55
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 41 | 55
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.135, Genalized Linear Mixed Models
Statistical Analysis 2: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.851, Generalized Linear Mixed Model

6. Secondary Outcome: Breastfeeding Self-Efficacy Scale
Description: Breastfeeding Self-Efficacy Scale is a 14 item scale with 5-point Likert scale (1-5). Score Range: 14-70, with higher scores (>50) indicate greater breastfeeding self-efficacy.
Time Frame: Baseline to 24 weeks
Population: The Breastfeeding Self-Efficacy Scale was completed each week by participants retained in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
score on a scale
  Baseline | 45.28 (13.71) | 45.49 (13.01)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 51.44 (13.48) | 51.26 (13.07)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 53.24 (14.04) | 51.62 (14.32)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 53.57 (14.07) | 51.90 (13.50)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 54.55 (14.84) | 54.10 (13.64)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 54.94 (14.94) | 54.91 (14.95)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 56.03 (14.54) | 55.13 (15.31)
  Week 18: number analyzed (Participants) | 73 | 128
  Week 18 | 57.24 (13.43) | 55.80 (15.63)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 54.31 (16.57) | 54.16 (16.23)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.571, Genalized Linear Mixed Models

7. Secondary Outcome: Anxiety Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form 6a
Description: The PROMIS Short Form v1.0 - Anxiety 6a is a 6-item Likert Scale (1-5, never - always). Total raw score range from 6-30. Raw scores are converted to a T-score. The T-score of 50 is the population mean and the average for the US population with a standard deviation of 10. The T-score of 60 is indicative of sub-clinical or elevated levels of anxiety. PROMIS Anxiety shows moderate to strong correlations with Generalized Anxiety Disorder 7-item scale and Hospital Anxiety and Depression Scale-Anxiety.
Time Frame: Baseline to 24 weeks
Population: Anxiety PROMIS measure was completed each week by participants retained in the study.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
T-score
  Baseline | 51.56 (9.10) | 51.27 (8.37)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 48.35 (8.71) | 49.81 (8.72)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 47.02 (8.29) | 48.36 (8.34)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 46.31 (7.55) | 48.49 (8.29)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 46.71 (7.62) | 46.58 (8.09)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 46.48 (8.31) | 46.54 (8.08)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 46.50 (7.90) | 47.45 (8.86)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 47.23 (8.59) | 47.23 (8.99)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 47.48 (8.79) | 47.63 (8.58)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.186, Genalized Linear Mixed Models

8. Secondary Outcome: Edinburgh Postnatal Depression Scale
Description: Edinburgh Postnatal Depression Scale is a 10-item questionnaire with a 0-3 Likert scale and a total score range from 0 to 30. A score of 10 or more may indicate possible depression and a score of 13 or higher may be used to identify women with higher depression levels.
Time Frame: Baseline to 24 weeks
Population: Edinburgh Postnatal Depression Scale was completed each week by participants retained in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
score on a scale
  Baseline | 5.56 (4.62) | 6.03 (4.92)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 4.56 (3.97) | 5.76 (4.32)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 4.05 (3.81) | 4.50 (3.84)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 3.15 (3.36) | 4.34 (4.13)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 3.45 (3.40) | 3.52 (3.75)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 2.84 (3.51) | 3.34 (3.75)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 3.00 (3.22) | 3.61 (4.00)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 3.42 (3.69) | 3.34 (3.57)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 4.22 (4.73) | 3.57 (3.91)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.191, Genalized Linear Mixed Models

9. Secondary Outcome: Fatigue Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form 6a
Description: The PROMIS Short Form v1.0 - Fatigue 6a is a 6-item Likert Scale (1-5, never - always). Total raw score ranges from 6-30. Raw scores are converted to a T-score. The T-score of 50 is the population mean and the average for the US population with a standard deviation of 10. The T-score of 60 is indicative of elevated levels of fatigue.
Time Frame: Baseline to 24 weeks
Population: Fatigue PROMIS measure was completed each week by participants retained in the study.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
T-score
  Baseline | 53.99 (9.63) | 54.95 (9.26)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 51.72 (10.62) | 54.48 (9.32)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 50.98 (10.25) | 52.26 (9.42)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 49.84 (9.89) | 52.59 (8.98)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 48.46 (10.01) | 50.46 (8.92)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 47.72 (9.56) | 49.81 (9.18)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 48.86 (9.82) | 48.82 (9.12)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 48.82 (9.61) | 49.53 (9.24)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 50.06 (10.03) | 50.24 (10.01)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.09, Genalized Linear Mixed Models

10. Secondary Outcome: Perceived Stress Scale10 Form V.09/16/13
Description: The Perceived Stress Scale (PSS-10) is a 10-item questionnaire is a 10-item Likert Scale from 0 ("Never") to 4 ("Very Often"). The total scores range from 0-40. To calculate a total PSS score, responses to the four positively stated items (items 4, 5, 7 and 8) first need to be reversed (i.e. 0 => 4; 1 => 3; 2 => 2; 3 => 1; 4 => 0). Higher scores indicate higher levels of perceived stress.
Time Frame: Baseline and 24 weeks
Population: Perceived Stress Scale measure was completed each week by participants retained in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
score on a scale
  Baseline | 12.94 (6.66) | 12.93 (6.15)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 11.52 (6.73) | 12.68 (6.26)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 10.71 (6.09) | 11.44 (6.30)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 9.51 (6.04) | 11.60 (6.05)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 10.33 (6.16) | 10.33 (6.03)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 10.10 (6.17) | 9.88 (6.17)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 10.52 (6.38) | 10.22 (6.19)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 11.15 (6.66) | 10.96 (6.09)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 11.39 (7.18) | 11.30 (6.70)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.672, Genalized Linear Mixed Models

11. Secondary Outcome: Sleep Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Sleep Disturbance 6a
Description: The PROMIS Short Form v1.0 - Sleep Disturbance 6a is a 6-item Likert Scale (1-5, never - always). Total raw score ranges from 6-30. Raw scores are converted to a T-score. The T-score of 50 is the population mean and the average for the US population with a standard deviation of 10. The T-score of 60 is indicative of increase sleep disturbances.
Time Frame: Baseline and 24 weeks
Population: Sleep PROMIS measure was completed each week by participants retained in the study.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | The BSM Intervention | Attention Control
Number analyzed (Participants) | 122 | 128
T-Score
  Baseline | 52.35 (9.16) | 54.13 (9.09)
  Week 1: number analyzed (Participants) | 108 | 116
  Week 1 | 49.32 (7.38) | 50.69 (8.45)
  Week 2: number analyzed (Participants) | 96 | 112
  Week 2 | 48.10 (6.96) | 48.91 (7.86)
  Week 3: number analyzed (Participants) | 94 | 107
  Week 3 | 47.44 (8.01) | 48.72 (8.24)
  Week 6: number analyzed (Participants) | 90 | 108
  Week 6 | 45.41 (7.51) | 47.79 (8.27)
  Week 9: number analyzed (Participants) | 81 | 99
  Week 9 | 45.65 (7.05) | 47.01 (8.57)
  Week 12: number analyzed (Participants) | 81 | 98
  Week 12 | 46.10 (7.07) | 47.61 (8.81)
  Week 18: number analyzed (Participants) | 73 | 93
  Week 18 | 47.99 (6.70) | 48.34 (8.66)
  Week 24: number analyzed (Participants) | 77 | 97
  Week 24 | 48.49 (8.81) | 47.70 (7.77)
Statistical Analysis 1: Comparison: The BSM Intervention vs Attention Control; Test type: Superiority; p = 0.221, Genalized Linear Mixed Models

ADVERSE EVENTS:
Time Frame: Baseline to 24 weeks
Description: Our definitions did not differ from the clinical trials.gov definitions.
Arm/Group | The BSM Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/128
Serious Adverse Events (participants affected / at risk) | 39/122 | 36/128
Other Adverse Events (participants affected / at risk) | 33/122 | 44/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The BSM Intervention (N=122) | Attention Control (N=128)
Preclampsia and Hypertension (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 7 (7) — Evaluation and hospital admission of hypertension preeclampsia
Urinary Tract Complications (Renal and urinary disorders) | 1 (1) | 2 (3) — Urinary track infections and procedures
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Cannabis reaction
Infections and Abscess (Infections and infestations) | 2 (2) | 1 (1) — Lip abscess, ingrown toenail, tooth pain
Musculoskeletal (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) — Injuries - hand, elbow, rib, motor vehicle accident
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) — Evaluations for Coronavirus disease 2019 (COVID-19) , colds, Streptococcus (Strep) throat, and respiratory flu
Mastitis and Nipple Infections (Reproductive system and breast disorders) | 5 (7) | 1 (1) — Infection of the breast and nipple with breastfeeding.
Heart Palpitations (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thyroid Evaluation and Surgery (Endocrine disorders) | 1 (2) | 3 (4) — Evaluation, admission, and or surgery of thyroid function
Infant Illness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) — Respiratory illness and tongue tie
Rash (Immune system disorders) | 1 (1) | 2 (3) — Rash and anaphylaxis
Abdominal Pain and Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 3 (3) — Assessment for abdominal pain and hemorrhoids
General illness and infections (Infections and infestations) | 3 (3) | 2 (2) — Malaise, fever
Sexual Transmitted Infections (Infections and infestations) | 2 (2) | 0 (0)
Birth Control Complications (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Postpartum Complications (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) — Spinal headache, bleeding, sciatic pain
Removal of Breast Mass (Surgical and medical procedures) | 1 (1) | 0 (0) — Preexisting to pregnancy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The BSM Intervention (N=122) | Attention Control (N=128)
Postnatal Depression (Pregnancy, puerperium and perinatal conditions) | 31 (57) | 40 (85) — Reported sum score of =/>10 on Edinburgh Postnatal Depression Scale (EPDS). A score of =/> 10 is indicative of clinical assessment for depression
Suicide Consideration (Psychiatric disorders) | 9 (13) | 14 (18) — EPDS #10 item asks if the participants has ideas of suicide or harm of themselves

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT05262920/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT05262920/ICF_001.pdf